CLINICAL TRIAL: NCT02530762
Title: A Randomized, Double-Blind, Crossover Study to Assess the Acute Gastrointestinal Tolerability Following a Single Serving of Cba-1, a Novel Dietary Fiber, in Healthy Men and Women
Brief Title: Acute Gastrointestinal Tolerability Following a Single Serving of a Novel Dietary Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: BIO-1409
Record Dates: First submitted 2015-08-20; First posted 2015-08-21 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Signs and Symptoms, Digestive
Keywords: Gastrointestinal tolerability; dietary fiber; clinical trial; healthy subjects
MeSH Terms: conditions — Signs and Symptoms, Digestive | interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Negative control (Placebo Comparator): No added fiber
  Interventions: Other: Negative Control
- Positive Fiber control (Active Comparator): 50g positive control fiber
  Interventions: Other: Positive Fiber control
- Novel Fiber 10g (Experimental): 10g novel fiber
  Interventions: Other: Novel Fiber
- Novel Fiber 30g (Experimental): 30g novel fiber
  Interventions: Other: Novel Fiber
- Novel Fiber 50g (Experimental): 50g novel fiber
  Interventions: Other: Novel Fiber

INTERVENTIONS:
Other: Novel Fiber — novel fiber supplemented beverage provided in one serving
  Other Names: Cba-1
  Arms: Novel Fiber 10g; Novel Fiber 30g; Novel Fiber 50g
Other: Positive Fiber control — positive control fiber supplemented beverage provided in one serving
  Other Names: Polydextrose
  Arms: Positive Fiber control
Other: Negative Control — No added fiber beverage
  Arms: Negative control

SUMMARY:
The study will assess the gastrointestinal tolerability of a single serving of a novel dietary fiber at three different dose levels in generally healthy men and women. Double-blind controlled, cross-over clinical trial with negative (no added fiber) and positive controls. Single dose, with 24 hours data collection and 1 week wash-out between cross-overs. 45 randomized, generally healthy men and women, 18-54 y, BMI higher or equal to 18.5 and smaller or equal to 39.99 kg/m2. Novel dietary fiber ingredient and positive control will be delivered in 240 ml beverages.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover study consisting of one screening visit (visit 1, day -7) and 10 test visits (days 0, 1, 7, 8, 14, 15, 21, 22, 28, 29). At the screening visit (visit 1, day -7), after subjects have provided informed consent, medical history and clinic visit procedures will be performed. Subjects who meet initial study inclusion/exclusion criteria will be instructed to maintain habitual diet and physical activity patterns throughout the study period. Subjects will also be instructed to avoid foods/beverages that cause Gastrointestinal (GI)-distress, as well as high-fiber foods for 24 h prior to the next clinic visit (visit 2, day 0). Additional instructions will include avoiding use of non-steroidal anti-inflammatory drugs (NSAIDS), antacids, proton pump inhibitors (PPIs), and H2 receptor antagonists for 24 h prior to the next clinic visit (visit 2, day 0).

At visit 2 (day 0), eligible subjects will return to the clinic following an overnight fast (9-14 h) to undergo clinic visit procedures. Adverse events (AEs) will also be assessed. Eligible subjects will then be randomly assigned to a test sequence wherein five test periods will be completed in a crossover design.

Subjects will be administered one serving of their assigned study product to be consumed in-clinic. Subjects will be instructed to consume the study product in its entirety within 15 min with a standard breakfast. Subjects will be dispensed a daily Bowel Habits Diary, which includes the Bristol Stool Scale, to record the frequency and consistency of bowel movements over the following 24 h (t = 0 is the time of study product consumption). Subjects will also be dispensed a 1-day diet record to record all foods/beverages consumed. Subjects will be instructed to record all foods/beverages for the following 24 h, beginning with study product consumption (t = 0 h). Subjects will be dismissed from the clinic with instructions to avoid foods/ beverages that cause GI-distress, as well as high-fiber foods, and to avoid use of non-steroidal anti-inflammatory drugs (NSAIDS), antacids, proton pump inhibitors (PPIs), and H2 receptor antagonists for the following 24 h until the next clinic visit (visit 3, day 1).

At visit 3 (day 1), subjects will arrive at the clinic 24 h after study product consumption following an overnight fast (9-14 h). Concomitant medication/supplement use, review of inclusion/exclusion, AEs will be assessed and subjects will complete a GI Tolerability Questionnaire. Subjects will also return their 1-day diet records and Bowel Habits Diary; this visit will be scheduled to ensure the entire 24 h period following study product consumption (t = 0 h) is captured. Prior to being dismissed from the clinic, subjects will be reminded of subsequent study visit instructions, including: fasting compliance (9-14 h, water only); maintenance of usual dietary and physical activity practices; avoiding use of non-steroidal anti-inflammatory drugs (NSAIDS), antacids, proton pump inhibitors (PPIs), and H2 receptor antagonists for 24 h prior to the next clinic visit (visit 4, day 7); and avoidance of foods/beverages that may cause GI distress, as well as high-fiber foods for 24 h prior to, and for the duration of the subsequent test visit (visit 4, day 7)].

Visit 2 procedures will be replicated at visits 4, 6, 8, and 10, which will be separated by a washout period of 7 ± 3 days. In addition, each subject will receive a copy of his or her 1-Day Diet Record from the first test visit (visit 2) and will be asked to replicate, as closely as possible, consumption of the same foods and to avoid foods/ beverages that cause GI-distress, as well as high-fiber foods. Visit 3 procedures will be replicated at visits 5, 7, 9, and 11.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18-54 years of age, inclusive.
* Subject has a body mass index (BMI) ≥18.50 and ≤39.99 kg/m2 at visit 1 (day -7) and has been weight stable (± 4.5 kg) for the previous 3 months.
* Subject is judged to be in good health on the basis of medical history.
* Subject is willing to maintain his or her habitual diet and physical activity patterns, including habitual use of study approved medications and/or dietary supplements throughout the study period.
* Subject is willing to avoid foods/beverages that cause GI-distress, as well as high-fiber foods for 24 h prior to, and following, visits 2, 4, 6, 8, and 10.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.

Exclusion Criteria:

* Subject reports any clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, history of surgery for weight loss, gastroparesis, and clinically important lactose intolerance).
* History or presence of clinically important endocrine (including type 1 or 2 diabetes mellitus), cardiovascular, pulmonary, biliary, renal, hepatic, pancreatic, or neurologic disorders that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
* Recent history (within 6 weeks of screening, visit 1) of constipation (defined as <3 bowel movements per week), and/or diarrhea (defined as ≥3 loose or liquid stools/d).
* Recent (within 6 weeks of screening, visit 1) episode of acute GI illness such as nausea, vomiting or diarrhea.
* Daily use of non-steroidal anti-inflammatory drugs (NSAIDS).
* Daily use of antacids, proton pump inhibitors, H2 blockers.
* Recent use of antibiotics (within 3 months of visit 2, day 0).
* Use of medications (over-the-counter and prescription) or dietary supplements (within 3 weeks of visit 2, day 0) known to influence GI function such as constipation medications and supplements (including laxatives, enemas, fiber supplements and/or suppositories); anti-diarrheal agents; anti-spasmodic; prebiotic and probiotic supplements.
* Extreme dietary habits, including but not limited to vegetarian diets and intentional consumption of a high fiber diet.
* Known allergy or sensitivity to food ingredients such as: soy, dairy (milk), wheat, egg, peanuts, tree nuts, fin fish and crustacean.
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg at visit 1, day -7). One re-test will be allowed on a separate day prior to visit 2 (day 0), for subjects whose blood pressure exceeds either of these cut points at visit 1, in the judgment of the Investigator.
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Any major trauma or surgical event within 2 months of visit 2, day 0.
* Females who are pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to use of a medically approved form of contraception throughout the study period. The method of birth control must be recorded in the source documentation.
* Exposure to any non-registered drug product within 30 days prior to the screening visit.
* Recent history of (within 12 months of visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Recent history of (within 2 months of visit 1) use of any tobacco-containing products.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, or confound the interpretation of the study results or put the subject at undue risk.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Composite gastrointestinal GI symptom score among conditions. | 24 hours
  Composite score will be calculated for each intake level as the sum of the ratings of the individual components (abdominal distention/bloating, gas/flatulence, borborygmus/stomach rumbling, and abdominal cramping). The ratings will be coded using a 4-point scale, in which 1 = none, 2 = mild, 3 = moderate, and 4 = severe.